CLINICAL TRIAL: NCT04072367
Title: A Prospective, Randomized, Open-Label, Multi-Center, Assessor-Blinded Study Designed to Compare the Safety, Performance and Efficacy of the NeVatm Stent Retriever Versus the Solitairetm Stent Retriever
Brief Title: FIrst-Pass Reperfusion With the NeVa Stent-Retriever Trial
Acronym: FIRST
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was withdrawn due to a change in company strategy.
Sponsor: Vesalio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VS-007
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2020-05

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Active Treatment Group (Other): NeVa Stent Retrievers
  Interventions: Device: NeVa Stent Retrievers
- Control Device (Other): Solitare Stent Retrievers
  Interventions: Device: Solitaire Stent Retrievers

INTERVENTIONS:
Device: NeVa Stent Retrievers — thrombus removal
  Arms: Active Treatment Group
Device: Solitaire Stent Retrievers — thrombus removal
  Arms: Control Device

SUMMARY:
This study is designed to compare the safety, performance and efficacy of blood clot (thrombus) removal in subjects presenting with acute ischemic stroke with the NeVa versus the Solitaire stent retrievers.

DETAILED DESCRIPTION:
A pivotal, randomized, open label, assessor-blinded, 90-day study designed to compare the safety, performance and efficacy of thrombus removal in subjects aged ≥ 18 years presenting with acute ischemic stroke with the NeVa versus the Solitaire stent retrievers.

A total of 414 eligible subjects will be randomized in a 1:1 ratio to one of two treatment groups:

* Active Treatment Group
* Control Device

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* A new focal disabling neurologic deficit consistent with acute cerebral ischemia
* NIHSS score ≥ 6;
* Prestroke mRS score of ≤ 2;
* Angiographic confirmation by DSA of an occlusion (eTICI 0-1) of the intracranial ICA, MCA-M1, MCA-M2, basilar artery, or intracranial vertebral artery with or without tandem involvement of the cervical ICA or cervical vertebral artery;
* Imaging Criteria:

  1. Strokes in the Anterior Circulation:

     * Non-Contrast CT (NCCT): ASPECTS 6 to 10 on baseline CT, or
     * CT perfusion (with Automated Volume Calculation): core infarct volume ≤ 70cc and Mismatch Ratio ≥ 1.5
     * CT perfusion (without Automated Volume Calculation): ASPECTS 6 to 10 on the CBV maps with Visualized MTT or TMax - CBV Mismatch greater than 50%, or
     * Brain MRI: ASPECTS 6 to 10 (and <70cc if Automated Volume Calculation is available) on baseline diffusion-weighted sequence (DWI).
  2. Strokes in the Posterior Circulation: pc-ASPECTS score 8 to 10 on baseline NCCT, CTA-source images, or DWI MRI.

     * Subjects for whom IV-tPA is indicated and who are available for treatment, are treated with IV-tPA within 4.5 hours of stroke onset (onset time is defined as the last time when the subject was witnessed to be at baseline), with verification that the subject has received/is receiving the correct IV t-PA dose for the estimated weight
     * Arterial puncture within 12 hours of symptom onset (or time last seen well - TLSW), thrombectomy procedure able to be completed within 2 hours from procedure start (arterial puncture).
     * Subject or legal representative is able and willing to give informed consent.

Exclusion Criteria:

* Rapid neurological improvement prior to groin puncture suggestive of resolution of stroke
* Seizures at stroke onset if it makes the diagnosis of stroke doubtful and precludes obtaining an accurate baseline NIHSS assessment.

  * Note: Subjects with a questionable seizure at onset of stroke should not be excluded if DSA confirms the presence of intracranial ICA and/or M1 occlusion, and accurate NIHSS can be obtained.
* Pre-existing medical neurological or psychiatric disease that would confound the neurological or functional evaluations, e.g. dementia with prescribed anti-cholinesterase inhibitor (e.g. Aricept).
* Cardiopulmonary resuscitation, significant cardiac arrhythmia, evidence of ongoing myocardial infarction, concern for pre-treatment pulmonary aspiration.
* Clinical symptoms suggestive of bilateral stroke or stroke in multiple territories.
* Cerebral vasculitis.
* History of severe allergy to contrast medium.
* Known allergy to stent retriever materials (nitinol, stainless steel);
* Suspicion of aortic dissection, septic embolus, or bacterial endocarditis.
* Active infection.
* Baseline CT or MRI showing mass effect or intracranial tumor (except small meningioma [≤ 3 cm]).
* CT or MRI evidence of recent/fresh hemorrhage on presentation.
* CTA, MRA, or DSA evidence of flow limiting carotid dissection, high-grade stenosis, or complete cervical carotid occlusion requiring stenting at the time of the index procedure (i.e., mechanical thrombectomy).
* Evidence of dissection in the intracranial cerebral arteries;
* Uncontrolled hypertension on presentation (defined as SBP > 220 mmHg and / or DBP > 120 mmHg). For subjects placed on intravenous BP medication, uncontrolled hypertension is defined as SBP > 185 mmHg and / or DBP > 110 mmHg.
* Baseline hemoglobin of < 7 mmol/L.
* Baseline platelet count < 50,000/uL.
* Renal failure as defined by a serum creatinine >3.0 mg/dL (264 mmol/L).

  * Note: subjects on renal dialysis may be treated regardless of serum creatinine levels.
* Known hemorrhagic diathesis, coagulation factor deficiency, or on anticoagulant therapy with INR > 3.0 or PTT > 3 times normal. Subjects on factor Xa inhibitor for 24-48 h ago must have a normal PTT.
* Baseline blood glucose of < 50 mg/dL (2.78 mmol) or > 400 mg/dL (22.20 mmol). Note: The ''correction'' of baseline glucose or coagulation laboratory values to meet inclusion criteria will not be allowed.
* Females who are pregnant or breastfeeding.
* Known current or recent use of illicit drugs or alcohol abuse.
* Use of an investigational drug or device within past 3 months;
* Life expectancy less than 6 months.
* Any other condition that, in the opinion of the investigator, precludes an endovascular procedure or poses a significant hazard to the subject if an endovascular procedure was performed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Reperfusion rate | post-procedure day 0
  The primary study endpoint is the reperfusion rate of the occluded target vessel (defined by an eTICI score ≥ 2b) following one single pass using the assigned stent retriever device(s)

SECONDARY OUTCOMES:
Stent retriever comparison | Day 90
  The secondary endpoint is the proportion of subjects treated with the NeVa device with good clinical outcomes at the Day 90 evaluation (defined as mRS score ≤ 2) when compared to the subjects treated with the predicate.

CONTACTS AND LOCATIONS:
Overall Officials: Raul Gomes Nogueira, MD, Principal Investigator — Emory University